CLINICAL TRIAL: NCT02563132
Title: Carbon Dioxide Insufflation Colonoscopy in Inflammatory Bowel Disease Patients
Brief Title: Carbon Dioxide Insufflation Colonoscopy in IBD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitkovice Hospital (Other)
Responsible Party: Principal Investigator, Premysl Falt, M.D., Ph.D., Premysl Falt, M.D., Ph.D., Vitkovice Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: DDC VN 08
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Colonoscopy; Carbon Dioxide; Inflammatory Bowel Disease
Keywords: colonoscopy; carbon dioxide; inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbon dioxide insufflation colonoscopy (CO2) (Experimental): Carbon dioxide during both insertion and withdrawal phase of the colonoscopy.
  Interventions: Procedure: Carbon dioxide insufflation
- Air insufflation colonoscopy (AI) (No Intervention): Air insufflation during both insertion and withdrawal phase of the colonoscopy.

INTERVENTIONS:
Procedure: Carbon dioxide insufflation — Carbon dioxide insufflation during diagnostic colonoscopy
  Arms: Carbon dioxide insufflation colonoscopy (CO2)

SUMMARY:
Carbon dioxide insufflation during colonoscopy significantly reduces discomfort (pain, bloating and flatulence) after the procedure. So far, it has not been studied in inflammatory bowel disease patients. The study was designed to evaluate discomfort after the carbon dioxide insufflation colonoscopy in comparison to standard air insufflation colonoscopy.

DETAILED DESCRIPTION:
Carbon dioxide insufflation during colonoscopy significantly reduces discomfort (pain, bloating and flatulence) during up to 24 hours after the procedure. So far, it has not been studied in inflammatory bowel disease patients who represent specific patient population indicated for colonoscopy. They are characterized by younger age, structural changes of the colon including intestinal resections and need for repeated and frequently difficult procedures.The study was designed to evaluate discomfort during 24 hours after the carbon dioxide insufflation colonoscopy in comparison to standard air insufflation colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* known diagnosis of Crohn´s disease and ulcerative colitis
* indication for diagnostic colonoscopy
* informed consent
* unsedated or minimally sedated procedure (< 3 mg of midazolam)

Exclusion Criteria:

* planned incomplete or therapeutic procedure
* deep sedation or general anesthesia
* intestinal resection longer than ileocecal resection
* isolated gastroduodenal or jejunal location of Crohn´s disease (L4)
* ulcerative proctitis (E1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Bloating score 1 hour after the colonoscopy | 1 hour
  Bloating severity on continuous scale 0-10 (0 = none, 10 = worst) 1 hour after colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Diseases Center - Vitkovice Hospital, Ostrava, Czechia